CLINICAL TRIAL: NCT03441958
Title: A Phase I-II Open-label Study of Reduced Intensity-allogeneic Transplant of ECT-001 (UM171/ Fed-batch Culture System) Expanded Cord Blood in Patients With High-risk Multiple Myeloma
Brief Title: ECT-001 (UM171) Expanded Cord Blood Transplant to Treat High-risk Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: ExCellThera inc. (Industry); Centre C3i (Unknown)
Responsible Party: Principal Investigator, Jean Roy, MD, Ciusss de L'Est de l'Île de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR007
Record Dates: First submitted 2018-02-02; First posted 2018-02-22 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
Keywords: hematopoietic stem cell transplant; Expanded cord blood
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECT-001 (UM171) expanded cord blood (Experimental): 1. Patients will receive a reduced intensity conditioning regimen containing Cyclophosphamide 50 mg/kg, Fludarabine 40 mg/m2 x 5 days and total body irradiation 200 cGy.
  2. The cord to be expanded is thawed 7 days prior to transplant and undergoes CD34+ selection. The CD34+ product will be placed in the fed-batch culture with UM171 for a 7-day expansion and is infused fresh on Day 0. The CD34- product is cryopreserved and will be thawed and infused on Day +1.
  3. Patients will receive standard supportive care and GVHD prophylaxis with Mycophenolate mofetil and Tacrolimus.
  Interventions: Biological: ECT-001 (UM171) expanded cord blood

INTERVENTIONS:
Biological: ECT-001 (UM171) expanded cord blood — ECT-001 expanded cord-blood will be produced and infused on site

SUMMARY:
Multiple Myeloma (MM) is a morbid disease associated with a poor outcome and while current therapies with new drugs have improved survival, MM still remains incurable in most patients. The only potential curative treatment remains allogeneic Hematopoietic stem cell transplant (HSCT), as shown by our cohort of 92 newly diagnosed patients who received a sibling tandem auto-allo (HSCT) with an estimated 10-year progression free survival (PFS) of 43%. However, the high incidences of toxicities including chronic graft-versus-host-disease (GVHD) (up to 79%) and disease progression (up to 49%) impair improvement in cure rate. Using umbilical cord blood (CB) as an alternative source of hematopoietic stem cells (HSC) could be superior biologically because of their increased proliferative capacity, greater number of progeny with longer telomeres and better anti-tumor efficacy in presence of positive residual disease. Moreover, using CB has been shown to decrease incidence of chronic GVHD. However, CBs have the disadvantage of having a limited HSC dose leading to prolonged cytopenia and higher risk of infections.

In a first in-human trial using CB expanded with the ECT-001 (UM171) molecule (clinicaltrial.gov # NCT02668315), the median net expansion of HSC was 36 fold, which allows for the selection of better HLA matched CB regardless of their lower HSC dose. Moreover, the ECT-001 expanded CBs have a different cell composition than regular CBs, with more than 25% of dendritic cell precursors. This, combined to better HLA matched CBs, may reduce chronic GVHD incidence and improve immune reconstitution. To date, 22 patients received an ECT-001 expanded CB and the procedure proved to be safe and feasible.

In this new trial, the goal is to evaluate the safety and efficacy of ECT-001 expanded CB transplant in high risk MM patients.

DETAILED DESCRIPTION:
This is a single institution, prospective, phase I/II open-label study in a maximum of 20 patients evaluating a novel treatment strategy in NDMM patients with high-risk disease who do not have a 6/6 compatible sibling donor. Participating patients will be from Hôpital Maisonneuve-Rosemont (HMR) or referred to HMR for this protocol. Newly diagnosed multiple myeloma patients will be evaluated for eligibility before or during the autologous stem cell transplant (ASCT) period. After a Bortezomib-based induction treatment (VTD, CyBorD, RVD or PAD [in patients with plasma cell leukemia]) for a minimum of 4 cycles, followed by Melphalan ≥ 140 mg/m2 and ASCT, eligible patients who accept to participate will undergo screening evaluation to receive a Reduced Intensity (RIC) allogeneic HSCT with ECT-001 expanded CB. It is estimated that 18 months will be necessary to enroll the targeted sample size.

Once eligibility has been confirmed, study treatment will begin. After an ASCT, eligible patients will receive a conditioning regimen before receiving a RIC allogeneic HSCT with an ECT-001 expanded CB on day 0. Patients will be followed at least every week for the first 3 months, then every month, in the absence of GVHD, for disease evaluation and adverse events. Occurrence and severity of acute GVHD will be evaluated using the modified Glucksberg176 and IBMTR177 criteria, while chronic GVHD will be evaluated using the NIH178 criteria.

The trial will be terminated when all patients have been followed for 5 years after allogeneic HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Newly diagnosed multiple myeloma using the International Myeloma Working Group criteria with measurable disease and any of the following:

   i. t(4;14), t(14;16), t(14;20), del(17p13), chromosome 1 abnormalities with ISS II or III; ii. Revised-ISS 3; iii. Primary plasma cell leukemia; iv. Refractory to first line triplet Bortezomib-based induction treatment. v. ≥ 2 cytogenetics abnormalities as defined above regardless of ISS stage
3. Received a first line triplet Bortezomib-induction regimen for a minimum of 4 cycles with achievement of at least partial response; or received a doublet or triplet Lenalidomide-based second line induction treatment with at least partial response for patients refractory to Bortezomib in first line.
4. Received high-dose Melphalan ≥ 140 mg/m2 followed by ASCT.
5. Availability of a cord blood with an HLA match ≥ 5/8 and < 8/8 meeting the following requirements: CD34+ cell count ≥ 0.5 x 105/kg and nucleated cell count >= 1.5 x 107/kg.

Exclusion Criteria:

1. Having previously received two ASCT.
2. Having previously received autologous-allogeneic tandem transplantation.
3. Having received more than 4 months of maintenance with Lenalidomide or Bortezomib after ASCT.
4. Poor organ function defined as either: forced vital capacity, forced expiratory volume in 1 second or lung diffusing capacity of carbon monoxide corrected for hemoglobin < 50%, left ventricular ejection fraction < 40% (evaluated by either echocardiogram or MUGA), uncontrolled arrhythmia or symptomatic cardiac disease, creatinine clearance < 60 mL/minute.
5. Karnofsky score < 70% or comorbidity index HCT-CI > 3.
6. Bilirubin > 2 x upper limit of normal (ULN) unless felt to be related to Gilbert's disease or hemolysis; AST and ALT > 2.5 x ULN; alkaline phosphatase > 5 x ULN; liver cirrhosis.
7. Non secretory disease or non-measurable disease in serum or urine at time of diagnosis.
8. Uncontrolled infection.
9. Active infection with any of the following viruses: HIV, HTLV-1 or 2, hepatitis B or C.
10. Presence of another malignancy with an expected survival estimated < 75% at 5 years.
11. Suspicion of cardiac amyloidosis.
12. Current history of drug and/or alcohol abuse.
13. Availability of a matched sibling donor.
14. Pregnancy, breastfeeding or unwillingness to use appropriate contraception.
15. Participation in a trial with an investigational agent within 30 days prior to entry in the study.
16. Patient unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up and tests.
17. Any abnormal condition or laboratory result that is considered by the principal investigator capable of altering patient's condition or study outcome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2025-10-17 (Estimated)

PRIMARY OUTCOMES:
Safety of ECT-001 expanded CB expansion as measured by toxicity evaluation | 5 years
  AEs with a CTCAE grade ≥ 3 (non hematologic) and with a grade ≥ 4 (hematologic) will be reported from the beginning of the conditioning regimen up to 5 years after CB transplant.
Feasibility of ECT-001 expanded CB expansion | 5 years
  Number of successful expansion and infusions in an outpatient nonmyeloablative transplant condition for high-risk myeloma patients
Measure of the kinetics of donor lymphoid cells recovery | 2 years
  Donor lymphocytes cells recovery assessed by chimerism analysis.
Measure of the kinetics of donor myeloid cells recovery | 2 years
  Time to neutrophils and platelets engraftment will be measured
Incidence of chronic GVHD by grade at 1 years by NIH criteria. | 1 year
  The incidence of chronic GVHD will be evaluated at 1 years using the recommendations of the NIH Consensus Conference and recently updated. Analysis by cumulative incidence
Incidence of chronic GVHD by grade at 2 years by NIH criteria. | 2 years
  The incidence of chronic GVHD will be evaluated at 1 years using the recommendations of the NIH Consensus Conference and recently updated. Analysis by cumulative incidence

SECONDARY OUTCOMES:
Correlation between neutrophil and CD34+ doses infused | 2 years
  Regression analysis
Correlation between neutrophil and CD34+CD45RA+ doses infused | 2 years
  Regression analysis. Time to neutrophil and platelet engraftment will be correlated to the CD34+ and the CD34+CD45RA- dose (which includes all human hematopoietic stem cells (HSCs): long term and short term repopulating cells) contained in the expanded graft. Expansion and cultures might change the characteristics and behaviour of CD34+ cells, hence the need to look at the correlation between primitive CD34+CD45RA- subpopulation and engraftment.
Incidence of graft failure | 2 years
  Cumulative incidence of graft failure by type (primary or secondary). For Primary engraftment failure will be defined as non-achieving a T lymphocyte chimerism of ≥30% at D+28 and ≥70% at D+180. Secondary graft failure will be defined as followed : ANC drops below 0.5x109/L for 14 consecutive days, unresponsive to G-CSF without any identifiable cause (medication, viral infection, vitamin deficiency or other) or <5% donor chimerism at any time point beyond initial engraftment in the absence of relapse and graft dominance by 2nd infused cord or other stem cell source.
Evaluation of T Cells reconstitution | 3 years
  Evaluation at several levels :
  * Multiparametric flow cytometry to quantify the proportion of naïve (CD45RA+/CD27+) and memory (CD45RA-/CD27+) cells.
  * TREC to measure thymic output
  * Diversity of the T cell repertoire (deep sequencing)
  * T-cell function (Elispot assays)
Evaluation of B cells reconstitution | 3 years
  B cell evaluation will be carried out prospectively using flow cytometry (CD19+), immunoglobulin (Ig) measurements, and PCR for donor B cell chimerism .
Evaluation of NK Cells reconstitution | 3 years
  NK cell evaluation will be performed by flow cytometry (CD 16+/56+) and chimerism analysis.
Evaluation of expanded HSC activity in vivo | 3 years
  Standard in vitro (long term culture-initiating cells and colony forming cells) and in vivo (the NSG mouse model) assays
Incidence of acute GVHD at day +120 | 4 months
  Analysis by cumulative incidence
Incidence of acute GVHD at 6 month | 6 months
  Analysis by cumulative incidence
Incidence of acute GVHD at 1 year | 1 year
  Analysis by cumulative incidence
Incidence of grade >=3 infectious complications | 5 years
  Analysis by cumulative incidence
Incidence of engraftment syndrome requiring therapy | 2 years
  Analysis by cumulative incidence
Duration of hospitalization | 6 months
  Number of days of hospitalization during the first 180 days post-transplant
Non relapse mortality at day +120 | 4 months
  Analysis by cumulative incidence
Non relapse mortality at 1 year | 1 year
  Analysis by cumulative incidence
Non relapse mortality at 2 year | 2 years
  Analysis by cumulative incidence
Progression free survival at 2 years | 2 years
  Kaplan Meier analysis
Overall survival at 2 years | 2 years
  Kaplan Meier analysis
Response to treatment at 1 year after allogeneic transplant | 1 years
  Evaluation of response categories according to the International Myeloma Working Group (IMWG)
Response to treatment at 2 year after allogeneic transplant | 2 years
  Evaluation of response categories according to the International Myeloma Working Group (IMWG)
Best response achieve at 1 year after allogeneic transplant | 1 years
  Evaluation of the best response during the 1 st year post-transplant
Best response achieve at 2 year after allogeneic transplant | 2 years
  Evaluation of the best response during the 2 years post-transplant
Minimal residual disease post transplant | 5 years
  Next Generation flow cytometry to determine how efficient an expanded CB is at reducing MM burden
Patient's quality of life | 5 years
  Assessment through Quality of Life questionnaires
Pharmaco-economic evaluation of the proposed treatment | 5 years
  Developement of an analysis model to determine if ECT-001 expanded CB to treat MM has a better cost-efficiency ratio than conventional chemotherapy-based treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean Roy, MD, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- CIUSSS de l'Est-de-l'île-de-Montréal, Installation Hôpital Maisonneuve Rosemond, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roy J, Cohen S, Sauvageau G, Ahmad I, Fournier V, Terra R, Caudrelier P, Thiant S, Thauvette G, Bambace N, Delisle JS, Lachance S, Kiss T, Bernard L, Roy DC, Veilleux O, LeBlanc R. A Pilot Study of UM171-Expanded Cord Blood Grafts for Tandem Auto/Allogeneic Hematopoietic Cell Transplant in High and Ultra-High-Risk Myeloma Patients. Transplant Cell Ther. 2025 Jan;31(1):34.e1-34.e14. doi: 10.1016/j.jtct.2024.10.008. Epub 2024 Oct 16. PMID 39419177